CLINICAL TRIAL: NCT00367276
Title: A Multicentre, Open, Uncontrolled Study to Assess Quality of Life During Six Cycles (24 Weeks) of Treatment With an Oral Contraceptive Containing 30 µg of Ethinylestradiol and 3 mg of Drospirenone (Yasmin).
Brief Title: Study to Evaluate the Effect of Six Cycles of Treatment With a Combined Oral Contraceptive (EE 0.30 mg/DRSP 3 mg) on Quality of Life.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91070; 305545
Record Dates: First submitted 2006-08-11; First posted 2006-08-22 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: Females requiring contraceptives
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination; drospirenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Yasmin (30 µg EE, 3 mg Drospirenone, BAY86-5131)

INTERVENTIONS:
Drug: Yasmin (30 µg EE, 3 mg Drospirenone, BAY86-5131) — Yasmin, SH T 470 FA; 30 µg ethinylestradiol and 3 mg drospirenone, oral administration over 6 treatment cycles, one tablet per day for 21 days followed by a 7 day pill-free interval.

SUMMARY:
The purpose of this study is to evaluate the effects on the quality of life and BMI of new contraceptives.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Female requiring contraceptives.
* Aged 18 to 35 if a non-smoker, aged 18 to 30 if a smoker.
* Regular menstrual cycle (defined as duration of 28 +/- 5 days).

Exclusion Criteria:

* No Contraindication for OC use

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2002-12; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Change of Psychological General Well Being Questionnaire score | pretreatment cycle to cycle 6

SECONDARY OUTCOMES:
Changes in body composition (evaluated by Multifrequency Bioelectrical Impedance Analysis) | pretreatment to cycle 6
Subject satisfaction with treatment at final visit | at final visit
Subject evaluation of changes in greasy skin and greasy hair | baseline to cycle 6

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer